CLINICAL TRIAL: NCT04920344
Title: Swallowing Outcomes and Circulating Tumor DNA in Patients With HPV Related Oropharyngeal Cancer Treated With Transoral Surgery and Reduced Intensity Adjuvant Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Matin Imanguli, MD, DDS, Assistant Professor. Chief of the Division of Head and Neck Surgical Oncology, Rutgers, The State University of New Jersey
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 032008; Pro2020002824 (Other: Rutgers Cancer Institute of New Jersey); NCI-2021-03006 (Registry Identifier: NCI CTRP registry); P30CA072720 (NIH)
Record Dates: First submitted 2021-06-02; First posted 2021-06-09 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Clinical Stage I HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Clinical Stage II HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Clinical Stage III HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Oropharyngeal Human Papillomavirus-Positive Squamous Cell Carcinoma
MeSH Terms: conditions — Oropharyngeal Neoplasms | interventions — Cisplatin; Circulating Tumor DNA; Physical Examination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- GROUP I - Low Risk Recurrence (transoral surgery, clinical observation)) (Active Comparator): After standard of care transoral surgery, patients whose small tumor was removed completely and have only one lymph node involved will undergo clinical observation.
  Interventions: Procedure: Transoral Surgery; Procedure: Incisional Tumor Biopsy; Other: Circulating tumor deoxyribonucleic acid (ctDNA) levels assessment; Other: MD Anderson Dysphagia Index; Other: University of Washington Quality of Life Questionnaire; Other: Euro-QOL 5 dimension scale questionnaire; Diagnostic Test: Modified barium swallow (MBS) evaluation with aspiration-penetration scale
- GROUP II - Medium Risk Recurrence (transoral surgery, EBRT 50Gy) (Experimental): Patients whose tumor was removed completely but has certain features that make it more likely to come back such as growth around the nerves or into the vessels, or has more than one lymph nodes involved, will undergo external body radiation therapy (EBRT) RT 50Gy for 5 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Transoral Surgery; Radiation: External Beam Radiation Therapy; Procedure: Incisional Tumor Biopsy; Other: Circulating tumor deoxyribonucleic acid (ctDNA) levels assessment; Other: MD Anderson Dysphagia Index; Other: University of Washington Quality of Life Questionnaire; Other: Euro-QOL 5 dimension scale questionnaire; Diagnostic Test: Modified barium swallow (MBS) evaluation with aspiration-penetration scale
- GROUP III - High Risk Recurrence (transoral surgery, EBRT 60Gy, cisplatin 30 mg/m2) (Experimental): Patients whose tumor has a "positive margin", which means the tumor could not be removed with healthy tissue around it or tumor grows significantly outside the lymph node will undergo EBRT RT 60 Gy for 6 weeks and receive cisplatin intravenously (IV) weekly 30mg/m2 for 6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Transoral Surgery; Radiation: External Beam Radiation Therapy; Drug: Cisplatin; Procedure: Incisional Tumor Biopsy; Other: Circulating tumor deoxyribonucleic acid (ctDNA) levels assessment; Other: MD Anderson Dysphagia Index; Other: University of Washington Quality of Life Questionnaire; Other: Euro-QOL 5 dimension scale questionnaire; Diagnostic Test: Modified barium swallow (MBS) evaluation with aspiration-penetration scale

INTERVENTIONS:
Procedure: Transoral Surgery — Patients will undergo transoral surgery
  Other Names: Therapeutic Conventional Surgery
Radiation: External Beam Radiation Therapy — Patients in Group II and Group III will undergo External Beam Radiation Therapy (EBRT) RT following transoral surgery.
  Other Names: EBRT
  Arms: GROUP II - Medium Risk Recurrence (transoral surgery, EBRT 50Gy); GROUP III - High Risk Recurrence (transoral surgery, EBRT 60Gy, cisplatin 30 mg/m2)
Drug: Cisplatin — Patients in Group III will receive cisplatin, 30 mg/m2, administered intravenously weekly per for 6 weeks.
  Other Names: Cisplatin Chemotherapy
  Arms: GROUP III - High Risk Recurrence (transoral surgery, EBRT 60Gy, cisplatin 30 mg/m2)
Procedure: Incisional Tumor Biopsy — Incisional biopsy of the primary tumor site will be required to confirm p16/HPV status of the tumor
Other: Circulating tumor deoxyribonucleic acid (ctDNA) levels assessment — Assess ctDNA levels at baseline, 2 weeks, 4 weeks, 10 weeks, 24 weeks and 1 year after the surgery.
  Other Names: Circulating ctDNA levels assessment
Other: MD Anderson Dysphagia Index — MDADI is a 20 item quality of life questionnaire specifically focusing on swallowing aspects. It was originally designed for head and neck cancer patients. The total score ranges from 20 to 100 with the higher score indicating higher level of function.
  Other Names: MDADI
Other: University of Washington Quality of Life Questionnaire — University of Washington Questionnaire is a 15 item quality of life instrument specifically designed for head and neck cancer patients.
  Other Names: UW QOL questionnaire
Other: Euro-QOL 5 dimension scale questionnaire — A generic quality of life and cost utility instrument widely used and validated for multiple disease settings, including head and neck cancer.
  Other Names: EQ-5D-5L
Diagnostic Test: Modified barium swallow (MBS) evaluation with aspiration-penetration scale — The videofluoroscopic modified barium swallow (MBS) study is the gold standard for for the evaluation of dysphagia, and specifically, airway protective mechanisms.
  The penetration/aspiration (PEN/ASP) scale is a routinely used eight-point scale designed to describe the depth of bolus penetration into the airway and the patient response to the penetration or aspiration.
  Other Names: MBS with PEN/ASP scale

SUMMARY:
This is a non-randomized, open-label phase II clinical trial that studies the effect of reduced dose radiation therapy and chemotherapy after surgery in treating patients with human papillomavirus (HPV) caused throat cancer. Giving reduced dose radiation therapy and chemotherapy after surgery may improve quality of life compared with standard of care primary chemoradiation approach without compromising survival.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To measure swallowing function and disease specific quality of life of patients with oropharyngeal cancer treated with transoral surgery and reduced intensity adjuvant therapy.

SECONDARY OBJECTIVES:

I. To examine kinetics of circulating tumor deoxyribonucleic acid (DNA) in patients treated with transoral surgery.

II. To estimate local control, progression free and overall survival using transoral surgery and reduced intensity adjuvant therapy.

OUTLINE: Based on pathologic findings after standard of care transoral surgery, patients are assigned to 1 of 3 groups.

GROUP I (LOW RISK): Patients whose small tumor was removed completely and have only one lymph node involved will undergo clinical observation.

GROUP II (MEDIUM RISK): Patients whose tumor was removed completely but has certain features that make it more likely to come back such as growth around the nerves or into the vessels, or has more than one lymph nodes involved, will undergo external body radiation therapy (EBRT) for 5 weeks in the absence of disease progression or unacceptable toxicity.

GROUP III (HIGH RISK): Patients whose tumor has a "positive margin", which means the tumor could not be removed with healthy tissue around it or tumor grows significantly outside the lymph node will undergo EBRT for 6 weeks and receive cisplatin intravenously (IV) weekly for 6 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven squamous cell carcinoma of the oropharynx
* Clinical stage T1-2, N0-N3, M0 by American Joint Committee on Cancer (AJCC) 8 criteria
* Must have tumors deemed surgically resectable with acceptable morbidity
* Estimated life expectancy of at least 12 weeks
* Must give informed consent
* Must have Eastern Cooperative Oncology Group (ECOG) performance status =< 3
* Must have detectable circulating HPV DNA levels
* Platelets >= 100,000/ul
* Absolute neutrophil count (ANC) >= 1,500/ul
* Hemoglobin > 8 g/dl (use of transfusion to achieve this is acceptable)
* Total bilirubin < 2 X institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) < 3 X institutional ULN
* Serum creatinine < 2 x institutional ULN or creatinine clearance > 50 ml/min as determined by 24 hour collection or estimated by Cockcroft-Gault formula
* Negative pregnancy test, if applicable

Exclusion Criteria:

* Patients may not have received previous therapy for their head and neck squamous cell carcinoma (SCC), including chemotherapy, radiation therapy, or surgery beyond biopsy
* Second primary malignancy. Exceptions are:

  * Patient had a second primary malignancy but has been treated and disease free for at least 3 years
  * In situ carcinoma (e.g. in situ carcinoma of the cervix)
  * Non-melanomatous carcinoma of the skin
* Patients with metastatic disease beyond the neck will be excluded
* Serious concomitant systemic disorders (including active infections) that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator
* Age < 18 years
* Patients with human immunodeficiency virus (HIV) infection are not automatically excluded, but must meet the following criteria: CD4 count is > 499/cu mm and their viral load is < 50 copies/ml. Use of highly active antiretroviral therapy (HAART) is allowed
* Grade 3-4 electrolyte abnormalities (Common Terminology Criteria for Adverse Events [CTCAE], version [v.] 5)

  * Serum calcium (ionized or adjusted for albumin) < 7 mg/dl (1.75 mmol/L) or > 12.5 mg/dl (> 3.1 mmol/L) despite intervention to normalize levels
  * Magnesium < 0.9 mg/dl (< 0.4 mmol/L) or > 3 mg/dl (> 1.23 mmol/L) despite intervention to normalize levels
  * Potassium < 3.0 mmol/L or > 6 mmol/L despite intervention to normalize levels
  * Sodium < 130 mmol/L or > 155 mmol/L despite intervention to normalize levels
* Women who are pregnant, due to the teratogenic effects of radiation therapy and chemotherapy on the unborn fetus. Women of childbearing age must agree to undergo a pregnancy test prior to therapy and to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and for 6 months after. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Tumor deemed unresectable with acceptable morbidity:

  * Tumors > 4 cm in size (T3 or higher)
  * Tumors of the base of tongue < 4 cm but with deep invasion of tongue musculature placing hypoglossal nerve or both lingual arteries at risk
  * Significant extension into hypopharynx
  * Extension into soft palate beyond 1/3 of the width
* Clinically extensive extranodal extension (ENE) e.g. radiologic evidence of invasion of carotid artery, gross extension into sternocleidomastoid muscle or deep neck muscles.

Lymph nodes larger than 6 cm without clinical ENE will be allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2025-05-08 (Estimated); Study Completion 2025-05-08 (Estimated)

PRIMARY OUTCOMES:
MD Anderson Dysphagia Index (MDADI) | At baseline.
  MDADI is a 20 item quality of life instrument specifically focusing on swallowing aspects. It was originally designed for head and neck cancer patients and has been widely used and validated in this population. The total score ranges from 20 to 100 with the higher score indicating higher level of function.
MD Anderson Dysphagia Index (MDADI) | At 24 weeks post completion of therapy.
  MDADI is a 20 item quality of life instrument specifically focusing on swallowing aspects. It was originally designed for head and neck cancer patients and has been widely used and validated in this population. The total score ranges from 20 to 100 with the higher score indicating higher level of function.
MD Anderson Dysphagia Index (MDADI) | At 1 year post completion of therapy.
  MDADI is a 20 item quality of life instrument specifically focusing on swallowing aspects. It was originally designed for head and neck cancer patients and has been widely used and validated in this population. The total score ranges from 20 to 100 with the higher score indicating higher level of function.

SECONDARY OUTCOMES:
Locoregional control. | At 3 years post completion of therapy
  Will be assessed using survival analysis (e.g., Kaplan-Meier method and Cox proportional hazards model).
Disease free survival. | At 3 years post completion of therapy
  Will be assessed using survival analysis (e.g., Kaplan-Meier method and Cox proportional hazards model).
Progression free survival. | At 3 years post completion of therapy
  Will be assessed using survival analysis (e.g., Kaplan-Meier method and Cox proportional hazards model).
Overall survival. | At 3 years post completion of therapy
  Will be assessed using survival analysis (e.g., Kaplan-Meier method and Cox proportional hazards model).
University of Washington Quality of Life Questionnaire | At baseline, 24 weeks and 1 year post completion of therapy
  University of Washington Questionnaire is a 15 item quality of life instrument specifically designed for head and neck cancer patients. Scoring is scaled to so that a score of 0 represents the worst possible response, and a score of 100 represents the best possible response. The higher the score - the better the outcome.
European Quality of Life Five Dimension Five Level Scale Questionnaire scores | At baseline, 24 weeks, and 1 year post completion of therapy
  Euro-QOL 5 dimension scale is a generic quality of life and cost utility instrument widely used and validated for multiple disease settings, including head and neck cancer.
  Euro-QOL 5 dimension scale is a preference-based HRQL measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The answers can be converted into EQ-5D index an utility scores anchored at 0 for death and 1 for perfect health. The EQ-5D questionnaire also includes a Visual Analog Scale (VAS), by which respondents can report their perceived health status with a grade ranging from 0 (the worst possible health status) to 100 (the best possible health status).
Rate of gastrostomy tube dependence | At baseline, 24 weeks, and 1 year post completion of therapy
  Percentage of patients requiring a gastrostomy tube after completion of therapy will be analyzed using generalized linear model (GLM) analysis.
Penetration-Aspiration Score on Modified Barium Swallow examination | Baseline and 1 year post completion of therapy
  Objective swallowing function assessment using modified barium swallow (MBS) evaluation with aspiration-penetration scale.
  The penetration/aspiration (PEN/ASP) scale is a routinely used eight-point scale designed to describe the depth of bolus penetration into the airway and the patient response to the penetration or aspiration. The higher the score, the worse is the outcome.
Correlation of circulating tumor deoxyribonucleic acid (ctDNA) levels with known adverse pathological features | At baseline and at 4 weeks post-surgery
  Correlation of ctDNA levels at baseline with known adverse pathological features such as, number of involved lymph nodes, extranodal extension and positive margins. Will be analyzed using GLM analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Matin Imanguli, MD, DDS, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (3):
- United States (3):
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - RWJBarnabas Health - Robert Wood Johnson University Hospital, New Brunswick, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey at University Hospital, Newark, New Jersey

IPD SHARING:
Plan to Share IPD: No